CLINICAL TRIAL: NCT04908319
Title: Hepatic Histopathology in Urea Cycle Disorders
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Lindsay Burrage, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-51257
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Urea Cycle Disorder; Ornithine Transcarbamylase Deficiency; Citrullinemia 1; ARGI Deficiency; ASL Deficiency; Argininosuccinic Aciduria; ASS Deficiency; Hyperargininemia; Carbamyl Phosphate Synthetase Deficiency; NAGS Deficiency
Keywords: Liver transplant; Liver disease; Liver biopsy; Histopathology
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Ornithine Carbamoyltransferase Deficiency Disease; Citrullinemia; Hyperargininemia; Argininosuccinic Aciduria; Carbamoyl-Phosphate Synthase I Deficiency Disease; N-acetyl glutamate synthetase deficiency; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Frozen liver samples, liver histology blocks/slides
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-site, retrospective chart review as well as a prospective study to evaluate histopathologic findings in liver samples from individuals with any UCD diagnosis. This study will be conducted at all Urea Cycle Disorders Consortium (UCDC) sites: Baylor College of Medicine in Houston, TX and Children's National Medical Center in Washington D.C.

DETAILED DESCRIPTION:
Urea cycle disorders (UCDs) are among the most common inborn errors of liver metabolism. With early diagnosis and improved treatments, the survival of individuals with UCDs has improved, and this improved survival has led to unmasking of some long-term complications such as hepatic dysfunction and progressive fibrosis in a subset of patients. Hepatic complications in UCDs are quite variable and dependent upon the specific metabolic defect.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary urea cycle disorder based on clinical suspicion confirmed by enzyme activity, DNA testing or metabolite analysis.
* History of liver transplantation and/or liver biopsy OR
* Planned liver transplantation and/or liver biopsy

Exclusion Criteria:

* Unavailability of histopathology report from the liver biopsy or explant, or unavailability of liver tissue or slides from the biopsy or explant OR
* Anticipated inability to obtain pathology report, liver disease, tissue blocks, or pathology slides after liver biopsy or transplantation
* Known history of a secondary cause for liver disease such as chronic viral hepatitis, autoimmune liver disease, short gut, small bowel syndrome, alcohol liver disease, or TPN-related cholestatic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with urea cycle disorders
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Hepatic fibrosis | Day 1
  Staging of fibrosis from histopathology report from the liver biopsy or explant
Steatosis | Day 1
  Grade of steatosis from histopathology report from the liver biopsy or explant
Hepatic glycogenosis | Day 1
  Presence and type of glycogenosis from histopathology report from the liver biopsy or explant

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Burrage, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Baylor College of Medicine, Houston, Texas